CLINICAL TRIAL: NCT07313540
Title: Feasibility of A Smartphone Application Intervention in Community Settings: A Pretest-Posttest Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-0082
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Aging; Dementia; Cognitive Decline
Keywords: Smarthphone; Tai-Chi; Meditation
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Twenty pairs of care recipients and caregivers (total: 40 people) will be recruited to the study and required to download the app to their phone and use it three times a week for four weeks. Tools to collect data include (1) one participation log, (2) two mood tests before and after the intervention, and (3) one feedback survey after the intervention.
  Interventions: Behavioral: utmbHealthyBrain Smartphone App

INTERVENTIONS:
Behavioral: utmbHealthyBrain Smartphone App — a wellness product related to relaxation and stress management and presents a low risk to the safety of users and other persons

SUMMARY:
The objective of this project is to test the feasibility of using a smartphone app in a community setting through collaborating with community-based organizations. The app is called utmbHealthyBrain and it has three activities: (1) drawing, (2) Tai-Chi and meditation, and (3) prayer reading. It also has a "share" function to enable users to interact with their family and friend. These activities can be translated to humans' well-beings such as a more stable emotion, more muscle movement, and better social engagement. This app does not collect any personal data and users are not required to register an account either. The overall study period is 6 weeks including one introduction session (week 1), four weeks of intervention (week 2 to 5), and final feedback session (week 6).

DETAILED DESCRIPTION:
This study will conduct primary data collection on 20 individuals aged 50+ and another 20 who are their caregivers regarding the use of a smartphone application (app) to promote mental well-being. The aging population is growing rapidly from 52 million in 2018 to 95 million by 2060. Approximately 34.2 million Americans have provided unpaid care to an adult age 50 or older. While 82% of them care for one adult, about 15% care for 2 adults and 3% for 3 or more adults. This number is expected to increase as the population ages. Deteriorating health of care recipients and caregivers is a critical issue that may be delayed by the use of a smartphone app to improve mental and emotional well-beings.

The objective of this proposed project is through collaborating with community-based organizations to test the acceptability and feasibility of a smartphone app intervention. We will collaborate with the community-based organization (i.e., UTMB OLLI and Libbie's Place) to announce the study by flyers and request RSVP to the study investigator. The investigator will provide instructions on using the smartphone app to potential participants and obtain participant's written consent to the study. After consenting, 20 pairs of older adults and their caregivers will fill out a mood test, download the app to their phone, and use it at least three times a week for four weeks. Participants will be required to keep their utilization log and fill out the post-intervention mood test and the feedback survey after four weeks of participation.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 50+ who has a primary source of assistance (no age limitation for the caregiver)
2. Both care recipient and caregiver can participate in the study for six weeks in total,
3. Both care recipient and caregiver can read, listen, write, and speak English
4. Both care recipient and caregiver have a personal smartphone.

Exclusion Criteria:

1. People who are diagnosed with any middle to severe cognitive symptoms (dementia or Alzheimer's Disease) or any psychiatric disease (depression, bipolar, PTSD, Schizophrenia, anxiety disorders, eating disorders)
2. People who are at hospice care
3. People who plan to move out of the current area in one year, and (4) people younger than 50 (but no age limitation for caregivers)

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a smartphone app intervention | 3 times per week for 4 weeks
  Feasibility will be assessed by participant adherence to the smartphone app intervention, defined as completion of activities three times per week.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chen Lee, PhD, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No